CLINICAL TRIAL: NCT03955874
Title: Practice Pattern Variation in Discontinuing Mechanical Ventilation in Critically Ill Adults: An International Prospective Observational Study
Brief Title: Mechanical Ventilation Discontinuation Practices
Acronym: IOS
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-024
Record Dates: First submitted 2019-05-03; First posted 2019-05-20 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Invasive Mechanical Ventilation; Critical Illness; Spontaneous Breathing Trial; Weaning Invasive Mechanical Ventilation; Tracheostomy; Direct Extubation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- INITIAL SBT: Patients who underwent an Spontaneous Breathing Trial prior to extubation. This cohort will be further subdivided into initial patients who initially pass an SBT successes and those who initially fail an SBT.
- DIRECT EXTUBATION: Patients that were directly extubated without conduct of a prior SBT or tracheostomy
- DIRECT TRACHEOSTOMY: Patients who underwent a direct tracheostomy without conduct of a prior SBT or extubation
- No attempt at mechanical ventilation discontinuation: Patients who died without conduct of a prior SBT, extubation or tracheostomy

SUMMARY:
Background: The requirement for ventilator support is a defining feature of critical illness. Weaning is the process during which the work of breathing is transferred from the ventilator back to the patient. Approximately 40% of the total time spent on ventilators is dedicated to weaning. The extent of practice variation in how this complex and expensive technology is discontinued from critically ill patients is unknown. Meanwhile, practice variation has been shown to adversely impact upon patient safety and clinical outcomes.

Purpose: To characterize practice pattern variation in weaning and the consequences of weaning variation by implementing an international, prospective observational study in Canada, the United States, the United Kingdom, Europe, India and Australia/New Zealand.

Primary Objectives: To describe

1. weaning practice variation among regions in 5 domains (the use of daily screening, preferred methods of support used before initial discontinuation attempts, use of written protocols, preferred methods of evaluating spontaneous breathing, and sedation and mobilization practices).
2. the assocation between selected discontinuation strategies and important clinical outcomes (length of stay, mortality, duration of ventilation).

Methods: The investigators propose to conduct a large scale, observational study involving critically ill adults requiring ventilator support for at least 24 hours to evaluate practices in discontinuing ventilators in 150 centres. The investigators will classify each new admission over the observation period according to the initial strategy that precipitated or facilitated ventilator discontinuation.

Relevance: This novel study will build collaborations with critical care investigators from around the world and industry

DETAILED DESCRIPTION:
Background: The requirement for mechanical ventilation is a defining feature of critical illness. Weaning is the process during which the work of breathing is transferred from the ventilator back to the patient. Approximately 40% of the total time spent on mechanical ventilation is dedicated to weaning. The extent and predictors of practice variation in how this complicated and expensive technology is discontinued from critically ill patients remains unknown. Meanwhile, practice pattern variability has been shown to adversely impact upon patient safety and important clinical outcomes.

Primary Objectives:

1. To describe weaning practice variation with regard to the (i) use of daily screening, (ii) preferred methods of support used before initial discontinuation attempts, (iii) use of written weaning and spontaneous breathing trial (SBT) protocols, (iv) preferred methods used to conduct SBTs and (v) sedation and mobilization practices among geographic regions.
2. To describe the association between variation in weaning practices (direct extubation, tracheostomy, SBT conduct) and important clinical outcomes.

   Secondary Objectives:
3. To identify baseline and time-dependent factors associated with use of selected strategies.
4. Among critically ill adults who undergo an initial SBT, the investigators will: a) investigate associations between SBT outcome (success/failure) and clinical outcomes, b) explore differences between critically ill patients who undergo an SBT early versus later in their intensive care unit (ICU) stay, and c) investigate the impact of different SBT techniques and humidification strategies on outcomes.
5. To identify important predictors (patient, clinician, SBT, institutional and regional) of SBT outcome.

Study Design and Population: The investigators propose to conduct an international prospective observational study of mechanical ventilation discontinuation practices in 150 ICUs involving all newly admitted critically ill adults requiring invasive ventilation for at least 24 hours.

Study Centres: Interested centres have been identified through completion of an information card enclosed in a previously administered International Weaning Survey. The investigators will use a multimodal approach to identify participating centers in each of the 6 geographic regions (Canada, the United States, the United Kingdom, Europe, India and Australia/New Zealand).

Study Outcomes: The investigators will classify each new admission over the study week according to the initial strategy that precipitated or facilitated mechanical ventilation discontinuation into one of five categories: direct extubation, tracheostomy, SBT success, SBT failure or death. The investigator will describe the association between the use of alternative discontinuation strategies and important clinical outcomes (e.g., mortality, ICU and hospital stay, ICU readmission and reintubation rates).

Relevance: Through collaborations with industry partners and international colleagues we will implement this large scale observational study to quantify the existence and extent of practice variation in weaning. Information obtained from this study will inform the design of future studies aimed at reducing weaning practice variation and improving outcomes in critically ill patients receiving invasive mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* All newly admitted critically ill adults after study initiation at participating ICUs.
* Requiring invasive mechanical ventilation for at least 24 (i.e. > or equal to 24) hours

Exclusion Criteria:

* Transferred to a participating ICU without a clear time of intubation
* Tracheotomy/tracheostomy present at the time of ICU admission
* Already on ventilator settings compatible with a SBT [e.g., T-piece or Continuous Positive Airway Pressure < or =5 cm H2O (water) or Pressure Support < or = 8 cm H2O (with or without PEEP) or Automatic Tube Compensation (ATC) or equivalent] at the time of ICU admission
* Patient residing in ICU for > or = 24 hours at the time of the study activation (i.e., not a new admission from the time of study activation).
* Patient readmitted to this ICU during the study period (i.e., would constitute a second inclusion) unless they were ineligible during their first admission
* Patients participating in studies (e.g., randomized controlled trials) with explicit weaning protocols incorporated into the study design

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We propose to conduct an International, Prospective Observational Study of Mechanical Ventilation Discontinuation Practices among critically ill adults who receive invasive mechanical ventilation for at least 24 (i.e., > or equal to 24) hours in approximately 150 international ICUs
Sampling Method: Non-Probability Sample
Enrollment: 1868 (Actual)
Dates: Start 2013-11-04 (Actual); Primary Completion 2016-12-17 (Actual); Study Completion 2016-12-17 (Actual)

PRIMARY OUTCOMES:
Practice variation among geographic regions in the use of daily screening to identify candidates to undergo an SBT | Through study completion (approximately 4 years)
  Use of once daily screening in clinical practice
Practice variation among geographic regions in the preferred methods of ventilator support used before initial discontinuation attempts | Through study completion (approximately 4 years)
  Differences in ventilator modes (Pressure Support, Assist Control, other) prior to discontinuation attempts
Practice variation among geographic regions in the use of written weaning and SBT protocols | Through study completion (approximately 4 years)
  Use of written protocols to liberate patients from ventilators
Practice variation among geographic regions in the methods used to conduct SBTs (and humidify oxygen) | Through study completion (approximately 4 years)
  Use of different techniques to conduct SBTs (Pressure Support, T-piece, etc.)
Practice variation among geographic regions in the sedation and mobilization practices during weaning | Through study completion (approximately 4 years)
  Use of different levels of sedation (Sedation Agitation Scale) and levels of mobilization (active, passive, none)
Association between variation in the weaning practices and total duration of ventilation. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and the total duration of ventilation.
Association between variation in the weaning practices and ICU mortality | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and ICU mortality.
Association between variation in the weaning practices and hospital mortality. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and hospital mortality.
Association between variation in the weaning practices and the proportion of patients off the ventilator at day 28. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and the proportion of patients off the ventilator at day 28.
Association between variation in the weaning practices and the proportion of patients out of the ICU at day 28. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and the proportion of patients out of the ICU at day 28.
Association between variation in the weaning practices and ICU LOS. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and ICU LOS (total and among survivors and non survivors).
Association between variation in the weaning practices and hospital LOS. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and hospital LOS (total and among survivors and non survivors).
Association between variation in the weaning practices and ICU readmission. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and ICU readmission (during the current hospitalization).
Association between variation in the weaning practices and reintubation. | Through study completion (approximately 4 years)
  We will describe the association between variation in the weaning practices and reintubation (or repeat ventilation following disconnection in tracheostomized patients) within 48 hours of extubation.

SECONDARY OUTCOMES:
Identify baseline characteristics and time-dependent factors associated with use of selected strategy (direct extubation, direct tracheostomy, Initial SBT) to discontinue mechanical ventilation | Through study completion (approximately 4 years)
  We will use cox proportion hazards modelling to identify baseline characteristics and time-dependent factors (development of adult respiratory distress syndrome, heart failure, acute kidney injury requiring dialysis) associated with the use of selected discontinuation strategies (direct extubation, direct tracheostomy, Initial SBT)
Association between initial SBT outcome (success/failure) and total duration of ventilation. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and the total duration of ventilation.
Association between initial SBT outcome (success/failure) and ICU mortality. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and ICU mortality.
Association between initial SBT outcome (success/failure) and hospital mortality. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and hospital mortality.
Association between initial SBT outcome (success/failure) and the proportion of patients off of the ventilator at day 28 | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and the proportion of patients off the ventilator at day 28.
Association between initial SBT outcome (success/failure) and the proportion of patients out of the ICU at day 28. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and the proportion of patients out of the ICU at day 28.
Association between initial SBT outcome (success/failure) and ICU LOS. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and ICU LOS (total and among survivors and non survivors.
Association between initial SBT outcome (success/failure) and hospital LOS. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and hospital LOS (total and among survivors and non survivors.
Association between initial SBT outcome (success/failure) and ICU readmission. | Through study completion (approximately 4 years)
  Association between initial SBT outcome (success/failure) and ICU readmission (during the current hospitalization).
Association between initial SBT outcome (success/failure) and reintubation. | Through study completion (approximately 4 years)
  Describe the associations between SBT outcome (success/failure) and reintubation (or repeat ventilation following disconnection in tracheostomized patients) within 48 hours of extubation
  c) Describe the association between different SBT techniques on clinical outcomes and d) Describe the association between use of selected humidification strategies and clinical outcomes.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on the total duration of ventilation. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the total duration of ventilation.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on ICU mortality. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU mortality.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on hospital mortality. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on hospital mortality.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on the proportion of patients off the ventilator at day 28. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the proportion of patients off the ventilator at day 28.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on the proportion of patients out of the ICU at day 28. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the proportion of patients out of the ICU at day 28.
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on ICU LOS. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU LOS (total and among survivors and non survivors).
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on hospital LOS. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on hospital LOS (total and among survivors and non survivors).
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on ICU readmission. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU readmission (during the current hospitalization).
Differences in clinical outcomes between patients who undergo an SBT early versus later in their ICU stay on reintubation. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on reintubation (or repeat ventilation following disconnection in tracheostomized patients) within 48 hours of extubation.
Association between different SBT techniques and total duration of ventilation. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the total duration of ventilation.
Association between different SBT techniques and ICU mortality. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU mortality.
Association between different SBT techniques and hospital mortality. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on hospital mortality.
Association between different SBT techniques and the proportion of patients off the ventilator at day 28. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the proportion of patients off the ventilator at day 28.
Association between different SBT techniques and the proportion of patients out of the ICU at day 28. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on the proportion of patients out of the ICU at day 28.
Association between different SBT techniques and ICU LOS. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU LOS (total and among survivors and non survivors).
Association between different SBT techniques and hospital LOS. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on hospital LOS (total and among survivors and non survivors).
Association between different SBT techniques and ICU readmission. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on ICU readmission (during the current hospitalization).
Association between different SBT techniques and reintubation. | Through study completion (approximately 4 years)
  Associations between use of different SBT technique (e.g., Pressure Support, T-piece) and the impact on reintubation (or repeat ventilation following disconnection in tracheostomized patients) within 48 hours of extubation
Association between use of selected humidification strategies and the total duration of ventilation. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on the total duration of ventilation.
Association between use of selected humidification strategies and ICU mortality. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on ICU mortality.
Association between use of selected humidification strategies and hospital mortality. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on hospital mortality.
Association between use of selected humidification strategies and the proportion of patients off the ventilator at day 28. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on the proportion of patients off the ventilator at day 28.
Association between use of selected humidification strategies and the proportion of patients out of the ICU at day 28. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on the proportion of patients out of the ICU at day 28.
Association between use of selected humidification strategies and ICU LOS. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on ICU LOS (total and among survivors and non survivors).
Association between use of selected humidification strategies and hospital LOS. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on hospital LOS (total and among survivors and non survivors).
Association between use of selected humidification strategies and ICU readmission. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on ICU readmission (during the current hospitalization).
Association between use of selected humidification strategies and reintubation. | Through study completion (approximately 4 years)
  Associations between use of different humidification strategies (e.g., Heat and Moisture Exchanger, heated humidifier) and the impact on reintubation (or repeat ventilation following disconnection in tracheostomized patients) within 48 hours of extubation.

OTHER OUTCOMES:
Predictors of initial SBT outcome. | Through study completion (approximately 4 years)
  Describe important predictors (patient, clinician, SBT, institutional and regional-related) of initial SBT outcome (SBT success and failure) using a single regression analysis. One analysis will be conducted to describe significant predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Karen E.A. Burns, MD, FRCPC, MSc, Principal Investigator — St. Michael's Hospital, Li Ka Shing Knowledge Institute, University of Toronto
Locations (14):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
- Canada (12):
  - Hamilton Health Sciences Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital Cancer Centre, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital Campus, London, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Hôpital Saint-Luc, Montreal, Quebec
  - Universite de Sherbrooke, Sherbrooke, Quebec
  - Universite Hopitalier de Sherbrooke, Sherbrooke, Quebec
  - Ciusss McQ, Trois-Rivières, Quebec

REFERENCES:
- [Background] Burns KEA, Rizvi L, Cook DJ, Lebovic G, Dodek P, Villar J, Slutsky AS, Jones A, Kapadia FN, Gattas DJ, Epstein SK, Pelosi P, Kefala K, Meade MO; Canadian Critical Care Trials Group. Ventilator Weaning and Discontinuation Practices for Critically Ill Patients. JAMA. 2021 Mar 23;325(12):1173-1184. doi: 10.1001/jama.2021.2384. PMID 33755077
- [Derived] Burns KEA, Rizvi L, Cook DJ, Dodek P, Slutsky AS, Jones A, Villar J, Kapadia FN, Gattas DJ, Epstein SK, Meade MO; Canadian Critical Care Trials Group. Variation in the practice of discontinuing mechanical ventilation in critically ill adults: study protocol for an international prospective observational study. BMJ Open. 2019 Sep 8;9(9):e031775. doi: 10.1136/bmjopen-2019-031775. PMID 31501132